CLINICAL TRIAL: NCT02674048
Title: Observational Study to Evaluate Clinical Practice and Satisfaction With Metvix® Daylight Photodynamic Therapy (PDT) in the Treatment of Mild and/or Moderate Actinic Keratosis of the Face and/or the Scalp
Brief Title: Metvix Daylight PDT in Actinic Keratosis
Acronym: SESAME
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: RD.03.SPR.104956
Record Dates: First submitted 2015-12-16; First posted 2016-02-04 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2017-01

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Metvix

SUMMARY:
Prospective non-interventional study conducted in Australia, Brazil, Mexico and Europe to evaluate clinical practice with Metvix Daylight PDT in the treatment of mild to moderate actinic keratosis of the face/scalp and to assess physician and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients to whom Metvix® Daylight-PDT has already been prescribed by their physician, according to the local label;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with mild to moderate Actinic Keratosis on the face or scalpe
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2015-09; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of physician satisfaction assessed on a 4-point scale from very satisfied to not satisfied with the question "Overall are you satisfied with Metvix DL-PDT?" | 3 months
Percentage of patient satisfisfaction assessed on a 4-point scale from very satisfied to not satisfied with the question "Overall, how satisfied are you with this treatment?". | 3 months

CONTACTS AND LOCATIONS:
Locations (7):
- See Jo-Ann, Sydney, New South Wales, Australia
- France, Pontoise, France
- Italy, L’Aquila, Italy
- Alkmaar, Alkmaar, Netherlands
- Madrid, Madrid, Spain
- Bern, Bern, Switzerland
- Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] See JA, Gebauer K, Wu JK, Manoharan S, Kerrouche N, Sullivan J. High Patient Satisfaction with Daylight-Activated Methyl Aminolevulinate Cream in the Treatment of Multiple Actinic Keratoses: Results of an Observational Study in Australia. Dermatol Ther (Heidelb). 2017 Dec;7(4):525-533. doi: 10.1007/s13555-017-0199-9. Epub 2017 Sep 13. PMID 28905294